CLINICAL TRIAL: NCT03458377
Title: Implementation of a Telephone Educational Intervention Performed in Outpatient Patients by the Gastrointestinal Endoscopy Nurse. Study of the Impact on the Pre-procedure, Procedure and Post-procedure Colonoscopy Quality Indicators.
Brief Title: Telephone Educational Intervention by the Gastrointestinal Endoscopy Nurse. Global Impact on the Quality of Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ESTRELLA
Record Dates: First submitted 2018-02-16; First posted 2018-03-08 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2018-02

CONDITIONS: Colonic Diseases; Nurse-Patient Relations; Educational Problems
Keywords: Colonoscopy; Quality; Telephone intervention
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Intervention Model Description: Reference population: all outpatient referred for the realization of a colonoscopy, regardless of the requesting Service.
  Two groups. One of them will receive an complete educational telephone call 7 days before de procedure in addition to the information received from the primary care center on the day of the request for the test. The inclusion in each one of the groups will be done through a randomization sheet.
  The intervention includes educational aspects:
  Explanation of the importance of making the test. Guidelines for the usual medication of the patient. Definition of fasting, explanation of colon cleansing adjusted to the presence of predictors of poor basic preparation. Explanation of the endoscopic procedure with the elimination of erroneous concepts of the patient with respect to the procedure. Explanation of norms of action subsequent to the endoscopy. Management of scheduling, destined to improve the adherence of the patient for the test.
Who Masked: Investigator
Masking Description: The endoscope that performs the colonoscopy and the person in charge of collecting the data of colonoscopy complications and the overall satisfaction of the procedure will be blind to the patient group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone call group (Experimental): The patient receives the colonoscopy information from the primary care center on the day of the request for the test and a 20 minute educational telephone call 7 days before de procedure.
  Interventions: Other: Educational telephone call
- Non-telephone call group (No Intervention): The patient only receives the colonoscopy information from the primary care center on the day of the request for the test.

INTERVENTIONS:
Other: Educational telephone call — Explanation of the importance of making the test. Guidelines for the usual medication of the patient. Definition of fasting, explanation of colon cleansing adjusted to the presence of predictors of poor basic preparation. Explanation of the endoscopic procedure with the elimination of erroneous concepts of the patient with respect to the procedure. Explanation of norms of action subsequent to the endoscopy. Management of scheduling, destined to improve the adherence of the patient for the test.
  Arms: Telephone call group

SUMMARY:
This study assesses what impact has on colonoscopy quality the implementation of a telephone educational intervention carried out individually on the patient in the days before the test. Half of the study patients will receive the educational intervention and the other half will not.

DETAILED DESCRIPTION:
A high-quality colonoscopy is an examination in with patients receive an indicated procedure, correct and relevant diagnoses are recognized or excluded, any therapy provided is appropriate, and all steps that minimize risk have been taken.

But quality also refers to pre-procedure and post-procedure quality issues such as information, booking, choice, privacy, dignity, aftercare and satisfaction of patients. All those issues can negatively affect the willingness of patients to perform the test and the possibility of preparing adequately. And what is more, it can diminish the quality of the own exploration, the satisfaction of the patients and their adherence to programs of endoscopic follow-up.

An action on these colonoscopy non-technical issues with a telephone educational intervention performed by the gastrointestinal endoscopy nurse can positively improve all (pre, intra and post-procedure) colonoscopy quality indicators.

ELIGIBILITY:
Inclusion Criteria:

* All outpatient referred from the Primary Care Centers to perform a colonoscopy in our Digestive Endoscopy Unit, regardless of the applicant's Service.

Exclusion Criteria:

* Hospital patients, patients who refuse inclusion in the study, patients included in another study, impossibility of carrying out the educational intervention and patients who are unable to obtain informed consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1534 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Colonoscopy non-adherence rate | At the moment of colonoscopy
  Ratio of patients do not attend the test

SECONDARY OUTCOMES:
Antiplatelet / anticoagulant rescheduling rate | At the moment of colonoscopy
  Ratio of patients attend the colonoscopy with poor adjustment of antiplatelet / anticoagulant medication so they need rescheduling of the test
Anesthetist rescheduling rate | At the moment of colonoscopy
  Ratio of patients attend the colonoscopy with American Society of Anesthesiologists (ASA) III / IV classification so they need rescheduling of the test under anesthesia
Bowel preparation rescheduling rate | At the moment of colonoscopy
  Ratio of patients attend the colonoscopy with inadequate Boston Bowel Preparation Scale (at least one of the colon segments with less than 2 points) so they need rescheduling of the test
Adenoma detection rate | At the moment of colonoscopy
  Ratio of patients with at least one adenoma in the colon
Cecal intubation rate | At the moment of colonoscopy
  Ratio of successful complete colonoscopies (cecal intubation or in case of previous surgery, ileocolic anastomosis)
Satisfaction of the endoscopic procedure | 30 days after colonoscopy
  Measurement of the overall satisfaction of the colonoscopy with a questionnaire validated by the American Society for Gastrointestinal Endoscopy (ASGE)
Complications related to colonoscopy | 30 days after colonoscopy
  Telephone interview. The patient will be asked about the appearance of perforation, hemorrhage and abdominal symptoms related to the test
Non-adequation colonoscopy cost of patient preparation for colonoscopy | From date of randomization until 30 days before colonoscopy
  Cost derived from non-adequation

CONTACTS AND LOCATIONS:
Overall Officials: Agustín Seoane Urgorri, MD, Principal Investigator — Parc de Salut Mar Hospital del Mar
Locations (1):
- Parc de Salut Mar. Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: SAP
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Access to the data will be available to the statistician of our institution.
URL: https://www.imim.es/sct/amib/amib.html

REFERENCES:
- [Background] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044
- [Background] Sola-vera J, Saez J, Laveda R, Girona E, Garcia-Sepulcre MF, Cuesta A, Vazquez N, Uceda F, Perez E, Sillero C. Factors associated with non-attendance at outpatient endoscopy. Scand J Gastroenterol. 2008;43(2):202-6. doi: 10.1080/00365520701562056. PMID 17852875
- [Background] Alvarez-Gonzalez MA, Flores-Le Roux JA, Seoane A, Pedro-Botet J, Carot L, Fernandez-Clotet A, Raga A, Pantaleon MA, Barranco L, Bory F, Lorenzo-Zuniga V. Efficacy of a multifactorial strategy for bowel preparation in diabetic patients undergoing colonoscopy: a randomized trial. Endoscopy. 2016 Nov;48(11):1003-1009. doi: 10.1055/s-0042-111320. Epub 2016 Aug 4. PMID 27490086